CLINICAL TRIAL: NCT03654547
Title: A Phase I, First-In-Human, Multicenter, Open-Label Study of TT-00420, Administered Orally in Adult Patients With Advanced Solid Tumors and Triple Negative Breast Cancers
Brief Title: Safety of TT-00420 (Tinengotinib) Monotherapy in Patients With Advanced Solid Tumors and Triple Negative Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TransThera Sciences (Nanjing), Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TT420X2101
Record Dates: First submitted 2018-08-21; First posted 2018-08-31 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumors; Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose Escalation arm followed by Dose Expansion arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation (Experimental): Eligible adult patients with advanced solid tumors will be enrolled into Dose Escalation cohorts and treated with TT-00420 at different dose cohorts. Starting dose will be 1 mg p.o., q.d. An ABLRM guided by the EWOC principle will evaluate the risk of under-dose or over-dose for the dose tested in each cohort and provide the recommendation dose for next cohort. Dose Escalation Teleconference will be held after the last evaluable patient complete Cycle 1 treatment in each dose cohort to evaluate DLT, determine MTD and/or DRDE.
  Interventions: Drug: TT-00420
- Dose Expansion (Experimental): A Dose Expansion cohort will be opened to enroll patients with selected advanced solid tumors and evaluate the safety, PK and preliminary efficacy of TT-00420 to determine the recommended phase 2 dose in patients with advanced solid tumors.
  Interventions: Drug: TT-00420

INTERVENTIONS:
Drug: TT-00420 — TT-00420 is an investigational, oral, multi-target, dual mechanism kinase inhibitor targeting both mitosis and tumor microenvironment, for the treatment of triple negative breast cancer (TNBC) and other advanced solid tumors.
  TT-00420 capsule will be administered once daily on a continuous schedule. A treatment cycle consists of 28 days.
  The proposed dosage form for early clinical research is powder filled hard gelatin capsule (PIC) with dosage strengths as of 1 mg, 5 mg and 20 mg.

SUMMARY:
This is a first-in-human, phase I clinical research study with TT-00420, an investigational, oral, multi-target, dual mechanism kinase inhibitor targeting both mitosis and tumor micro-environment, for the treatment of triple negative breast cancer (TNBC) and other advanced solid tumors. The study consists of a dose escalation part followed by a MTD expansion part.

DETAILED DESCRIPTION:
Dose Escalation Cohorts: Eligible adult patients with advanced solid tumors will be enrolled into Dose Escalation cohorts. Starting dose of TT-00420 mono-therapy will be 1 mg p.o., q.d. TT-00420 capsule will be administered once daily on a continuous schedule. A treatment cycle consists of 28 days. An ABLRM guided by the EWOC principle will evaluate the risk of under-dose or over-dose for the dose tested in each cohort and provide the recommendation dose for next cohort. Dose limiting toxicity (DLT) will be evaluated per the pre-defined DLT criteria and managed by the pre-defined rules detailed in the protocol. Maximum Tolerated Dose (MTD) and/or Dose Recommend for Dose Expansion (DRDE) will be determined in Dose Escalation cohorts.

Dose Expansion Cohorts:

TNBC Cohort:

TNBC Dose-Expansion cohort will be opened to enroll the patients with advanced TNBC and evaluate the safety, PK and preliminary efficacy of TT-00420 to identify the optimal biological dose (OBD), when feasible, in patients with advanced TNBC.

SAT Cohort:

A parallel basket SAT Dose Expansion Cohort will be open to enroll patients with selected advanced tumors (SAT) to evaluate the safety, PK and preliminary efficacy of TT-00420 to identify the optimal biological dose (OBD), when feasible, in patients with SATs.

Recruitment in dose expansion cohorts may be put on hold if any significant safety finding(s) that was not observed in dose escalation cohorts is identified. Bayesian modeling will be updated with the new findings to evaluate if the previously determined MTD or DRDE still suitable for further enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years to 75 years at the time of provision of informed consent
2. Dose Escalation Cohorts: Histopathological or cytologically documented locally advanced or metastatic solid tumors who have no available standard therapeutic treatment options Dose Expansion Cohorts: Histopathological or cytologically documented locally advanced or metastatic TNBC or SATs
3. TNBC Dose Expansion Cohort:

   1. Histologically proven invasive breast carcinoma with triple negative receptor status per institutional standard and with confirmed negative for ER and PR by IHC (<10% positive tumor nuclei)
   2. relapsed/refractory to at least one line of systemic chemotherapy
4. At least one measurable lesion as defined by RECIST V1.1 criteria for solid tumors
5. ECOG performance status of 0 or 1
6. Adequate organ function confirmed at Screening and within 10 days of initiating treatment, as evidenced by:

   * Absolute Neutrophil Count (ANC) ≥ 1.5 x 10^9/L
   * Hemoglobin (Hgb) ≥ 9 g/dl
   * Platelets (plt) ≥ 100 x 10^9/L
   * AST/SGOT and ALT/SGPT ≤ 2.5 x Upper Limit of Normal (ULN) or ≤ 5.0 x ULN if liver metastases are present
   * Total bilirubin ≤ 1.5 x ULN, or direct bilirubin < ULN for patients with total bilirubin levels >1.5 ULN
   * Serum creatinine ≤ 1.5 x ULN or calculated 24-hour clearance ≥ 50 mL/min
   * Negative pregnancy test within 72 hours before starting study treatment in all pre-menopausal women and women < 12 months after the onset of menopause
7. Must agree to take sufficient contraceptive methods to avoid pregnancy during the study and until at least 6 months after ceasing study treatment
8. Able to sign informed consent and to comply with the protocol

Exclusion Criteria:

1. Women who are pregnant or lactating
2. Women of child-bearing potential (WOCBP) who does not use adequate birth control
3. Patients with any hematologic malignancy. This includes leukemia (any form), lymphoma, and multiple myeloma.
4. Patients with

   1. a history of primary central nervous system tumors or
   2. carcinomatous meningitis Note: Patients with treated brain metastases that are off corticosteroid and have been clinically stable 28 days are eligible for enrollment
5. Patients with the following mood disorders as judged by the Investigator or a psychiatrist, or as result of patient's mood assessment questionnaire:

   * Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia; a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others)
   * ≥ CTCAE grade 3 anxiety
   * The psychiatric judgment, if available, overrules the mood assessment questionnaire result/investigator judgment
6. Impaired cardiac function or clinically significant cardiac diseases, including but not limited to any of the following:

   1. LVEF < 45% as determined by MUGA scan or ECHO
   2. Congenital long QT syndrome
   3. QTc ≥ 450 msec on screening ECG
   4. Unstable angina pectoris ≤ 3 months prior to starting study drug
   5. Acute myocardial infarction ≤ 3 months prior to starting study drug
7. Patients with

   1. unresolved diarrhea ≥ CTCAE grade 2, or
   2. impairment of gastrointestinal (GI) function, or
   3. GI disease that may significantly alter the absorption of TT-00420 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
8. Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., uncontrolled hypertriglyceridemia [triglycerides > 500 mg/dL], active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol
9. Patients who have received chemotherapy, targeted therapy or immunotherapy ≤ 4 weeks (6 weeks for nitrosourea or mitomycin-C) prior to starting study drug or who have not recovered from side effects of such therapy
10. Patients who have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
11. Patients who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
12. Patients who have been treated with any hematopoietic colony-stimulating growth factors (e.g., G-CSF, GM-CSF) ≤ 2 weeks prior to starting study drug. Erythropoietin or darbepoetin therapy, if initiated before enrollment, may be continued
13. Patients who are currently receiving treatment with therapeutic doses of warfarin sodium (Coumadin®) or any other coumarin-derivative anticoagulants
14. Patients who have received corticosteroids ≤ 2 weeks prior to starting study drug or who have not recovered from the side effects of such treatment
15. Patients who are currently receiving treatment with medication that has known risk to prolong the QT interval or inducing Torsades de Pointes, and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug
16. Patients who are receiving high to moderate CYP3A inhibitors and inducers as listed in Appendix F
17. Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory)
18. Known history of active infection with Hepatitis B (e.g., HBsAg reactive), or Hepatitis C (e.g., HCV RNA (qualitative) is detected)
19. Has received a live-virus vaccination within 30 days of planned first dose Note: Seasonal flu vaccines are permitted.
20. Inability to swallow or tolerate oral medication
21. Has a history or current evidence of any condition, therapy, or laboratory abnormality that, in the opinion of the investigator, might confound the results of the trial, interfere with the patient's participation and compliance in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and/or Dose Limiting Toxicity (DLT) | At the end of Cycle 1 (each cycle is 28 days)
  FIH Dose Finding

SECONDARY OUTCOMES:
Dose Recommended for Dose Expansion (DRDE) | At the end of Cycle 1 (each cycle is 28 days)
  Dose Recommended for Dose Expansion
Optimal Biological Dose (OBD) | At the end of Cycle 1 (each cycle is 28 days)
  Dose Recommended for Dose Expansion
Number of Participants With Abnormal Laboratory Values | Up to 30 days from study discontinuation
  Safety and tolerability of TT-00420
Number of Participants With Adverse Events That Are Related to Treatment | Up to 30 days from study discontinuation
  Safety and tolerability of TT-00420
Peak Plasma Concentration (Cmax) of TT-00420 | through study completion, an average of 6 months
  PK parameters of TT-00420
Time at which Cmax was first observed (Tmax) of TT-00420 | through study completion, an average of 6 months
  PK parameters of TT-00420
Half-life (T1/2) of TT-00420 | through study completion, an average of 6 months
  PK parameters of TT-00420
Objective Response Rate (ORR) | through study completion, an average of 1 year
  ORR of TT-00420 in patients with TNBC or SAT treated in Dose Expansion cohorts
Disease Control Rate (DCR) | through study completion, an average of 1 year
  DCR of TT-00420 in patients with TNBC or SAT treated in Dose Expansion cohorts
Duration of Response (DOR) | through study completion, an average of 1 year
  DOR of TT-00420 in patients with TNBC or SAT treated in Dose Expansion cohorts
Progression Free Survival (PFS) | through study completion, an average of 1 year
  PFS of TT-00420 in patients with TNBC or SAT treated in Dose Expansion cohorts
Overall Survival (OS) | through study completion, an average of 1 year
  OS of TT-00420 in patients with TNBC or SAT treated in Dose Expansion cohorts

OTHER OUTCOMES:
Exploratory Biomarker Assay | through study completion, an average of 6 months
  TNBC subtype; pH3, angiogenesis, p-STAT3 etc.; MSI, TMB

CONTACTS AND LOCATIONS:
Overall Officials: Sarina A. Piha-Paul, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- MD Anderson Cancer Center, Houston, Texas, United States
- Cancer Hopital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peng P, Qiang X, Li G, Li L, Ni S, Yu Q, Sourd L, Marangoni E, Hu C, Wang D, Wu D, Wu F. Tinengotinib (TT-00420), a Novel Spectrum-Selective Small-Molecule Kinase Inhibitor, Is Highly Active Against Triple-Negative Breast Cancer. Mol Cancer Ther. 2023 Feb 1;22(2):205-214. doi: 10.1158/1535-7163.MCT-22-0012. PMID 36223547